CLINICAL TRIAL: NCT03287427
Title: First-in-human Phase I Clinical Trial of a Combined Immune Modulatory Approach Using TetMYB Vaccine and Anti-PD1 Antibody in Patients With Advanced Solid Cancer Including Colorectal or Adenoid Cystic Carcinoma.
Brief Title: MYPHISMO: MYB and PD-1 Immunotherapies Against Multiple Oncologies Trial
Acronym: MYPHISMO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYPHISMO
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer; Adenoid Cystic Carcinoma
Keywords: Advanced; Metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Adenoid Cystic; Neoplasm Metastasis | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TetMYB Vaccine & BGB-A317 (Experimental)
  Interventions: Drug: TetMYB Vaccine; Drug: BGB-A317

INTERVENTIONS:
Drug: TetMYB Vaccine — Weekly intra-dermal injections of either 0.1mg, 0.5mg or 1.0mg on day 1 for week 1 to week 6.
Drug: BGB-A317 — 3 weekly IV injections of 200mg commencing from Week 4.

SUMMARY:
The purpose of this research study is to look at the effects, good or bad, of TetMYB Vaccine in combination with BGB-A317 in patients with advanced or metastatic solid cancers (including colorectal or adenoid cystic cancer).

The immune system is the body's defence against cancer, bacteria and viruses. TetMYB Vaccine is a vaccine that helps your immune system to recognise the cancer cells. BGB-A317 is an antibody (a type of protein made in the body in response to a foreign substance) that helps to stop or reverse the growth of tumour cells.

Up to 32 participants may take part in this study, which is divided into 2 stages: dose escalation (different doses will be tested in small groups of patients) and dose expansion (one or more doses may be tested in a larger group of patients). Which stage you participate in will depend on which is open at the time. Your study doctor will discuss this with you.

During dose escalation, study patients will receive increasing doses of the TetMYB Vaccine, starting at a low dose. During dose expansion, study patients will receive the dose determined as safe in dose escalation.

The study design is as follows:

In the dose finding stage, the first patient of each dose level will receive 6 consecutive weekly doses of intradermal TetMYB monotherapy for safety evaluation. If there are no reported DLTs, the next 2 patients of the same dose level will also receive 6 consecutive weekly intradermal doses of TetMYB, however with 3 weekly doses of BGB-A317 commencing with the fourth TetMYB dose. The dosage of TetMYB are as follows:

* Dose level 1: 100 ug in 100 uL of sterile dH2O containing 5% DMSO
* Dose level 2: 500 ug in 100 uL of sterile dH2O containing 5% DMSO
* Dose level 3: 1000 ug in 100 uL of sterile dH2O containing 5% DMSO.

In the dose expansion stage, the dosage will be the maximum tolerated dose (MTD) identified in the dose-finding stage and in combination with BGB-A317.

TetMYB Vaccine is being developed and manufactured by the Peter MacCallum Cancer Centre according to Good Manufacturing Practice (GMP) and in accordance with guidelines provided by the Food and Drug Administration (FDA) in the USA and Therapeutic Goods Administration (TGA) in Australia. TetMYB Vaccine is an experimental treatment and is currently not approved for use in any country. This means that it is not an approved treatment for cancer in Australia. This will be the first time that the TetMYB vaccine is given to humans.

BGB-A317 is being developed by BeiGene, a biopharmaceutical company. BGB-A317 is an experimental treatment. This means that it is not an approved treatment for solid cancers in Australia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years or older at screening.
2. Patients with advanced/metastatic colorectal or adenoid cystic carcinoma; for which no effective standard therapy is available.
3. Patient has been fully informed about the study and is willing to participate in the study, and has provided written informed consent prior to any trial specific screening procedures.
4. Measurable disease as per irRECIST criteria 1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
6. Life expectancy greater than 3 months.
7. Adequate haematological, renal and hepatic functions as defined by:

   * Neutrophil count >1.5 x 109/L
   * Platelets >100 x 109/L
   * Hb >100 g/L (Patients can be transfused in the lead-in period, providing they do not have active bleeding or require regular transfusions)
   * Total bilirubin <1.5x upper limit of normal (ULN)
   * ALT and AST <2.5x ULN (<5.0x ULN for patients with hepatic metastasis)
   * Serum creatinine <1.5x ULN or Creatinine Clearance >50 mL/min (Cockcroft-Gault or Nuclear GFR method)
8. Willing to provide study specific pre-treatment biopsy of tumour and allow use of archival tumour biopsies. This is optional for adenoid cystic carcinoma patients.
9. Willing to consent to the use of their collected fresh tumour and archival FFPE specimen and blood samples as detailed in the protocol for research including but not limited to DNA, RNA and protein based biomarker detection.
10. Men and women of childbearing potential must use adequate contraception to prevent pregnancy during the study. Adequate contraception is defined in the study as any medically recommended method (or combination of methods) as per standard of care. An adequate contraception includes hormonal contraception with implants or combined oral, transdermal or injectable contraceptives, certain intrauterine devices, bilateral tubal ligation, hysterectomy, or vasectomy of partner. Combinations of male condom with either cap, diaphragm or sponge with spermicide are also considered acceptable. For women of childbearing age, a negative pregnancy test needs to be confirmed before inclusion.

Exclusion Criteria:

1. Prior therapy with an anti-cancer vaccine; or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
2. Chemotherapy, radioactive, biological cancer therapy, or tyrosine kinase inhibitor (TKI) therapy, within four weeks prior to the first dose of study drug. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE v4.03) or baseline before administration of study drug.
3. Patient has had a prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, or localized prostate cancer.
4. Uncontrolled or significant intercurrent or recent illness including:

   * Autoimmune disorder or history of autoimmune disease requiring immunosuppressive treatment
   * Cardiac disorder such as uncontrolled cardiac failure, unstable angina or non-ST segment elevation myocardial infarction (NSTEMI) or myocardial infarction, uncontrolled arrhythmia less than 3 months before screening
   * Active or uncontrolled severe infection
5. History of solid organ transplantation or any condition requiring chronic treatment with corticosteroids or other immunosuppressive agents.
6. Active coagulopathy/bleeding diathesis.
7. Cirrhosis, chronic active or untreated persistent hepatitis.
8. Active Hepatitis B: (defined as having a positive Hepatitis B surface antigen [HBsAg] test at screening). Patients with past or resolved Hepatitis B infection (defined as having a negative HBsAg test and a positive IgG antibody to Hepatitis B core antigen [anti-HBc]) are eligible. Hepatitis B virus (HBV) DNA must be obtained in these patients prior to Cycle 1, Day 1, and must demonstrate no active infection.
9. Active Hepatitis C: Patients positive for Hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
10. History of adverse reactions to peptide vaccines.
11. Patients who are pregnant or lactating.
12. Has received an investigational drug within 4 weeks prior to first dose of study drug, or unless other has been agreed with the SSC.
13. Is currently receiving any agent with a known effect on the immune system, unless at dose levels that is not immunosuppressive (e.g. prednisone at 10 mg/day or less or as inhaled steroid at doses used for the treatment of asthma).
14. Known history of positive tests for HIV/AIDS.
15. Prior treated brain metastases must be without evidence of progression (through magnetic resonance imaging [MRI] with contrast - preferred method or contrast enhanced computed tomography [CT]) for at least 4 weeks and off immunosuppressive doses of systemic medications, such as steroids (doses > 10 mg/day prednisone or equivalent) for at least 2 weeks before study drug administration to be eligible
16. Receipt of live, attenuated vaccine within 28 days prior to the first dose of study drug (Note: Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of study drug).
17. Any contraindication to receiving anti-PD-1 antibody (BGB-A317) or hypersensitivity to the constituents of BGB-A317.
18. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
19. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
The incidence of Grade 3 or 4 or greater adverse events (AEs) according to CTCAE v4.03 criteria and clinical laboratory abnormalities defined as dose-limiting toxicities (DLTs). | End of Week 6

SECONDARY OUTCOMES:
Tolerability of the treatment as defined as receiving a minimum of 4 doses of TetMYB Vaccine within 6 weeks of starting treatment. | End of Week 6
The occurrence, type, severity and relationship to treatment of adverse events occurring after the first 6 weeks of treatment, described according to CTCAE v4.03 criteria. | Week 7 and through study completion, an average of 12 months.
The objective response as defined by the achievement of a complete (irCR) or partial (irPR) response, based on irRECIST criteria within 12 weeks of first vaccination. | End of Week 12
Clinical benefit as defined by wither the achievement of a complete (irCR) or partial (irPR) response as per irRECIST criteria; or the maintenance of stable disease (irSD), as per irRECIST criteria, at 12 weeks after commencement of treatment. | End of Week 12.
Progression free survival (PFS) as defined as the time from first vaccination to the earliest of date of disease progression as assessed by irRECIST or death from any cause. | From the date of treatment commencement to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
Overall survival (OS) as defined as the time from first vaccination to date of death from any cause. | From the date of treatment commencement to the date of death from any cause, whichever came first, assessed up to 48 months..
To demonstrate a MYB-specific immune response through epitope stimulation of PBMCs and assessment with CBA, FACS for IFN-γ and TNF-α production, and via the evaluation of changes in tumour microenvironment in pre- and post-treatment biopsies. | Through study completion, an average of 48 months.
To assess metabolic response, as assessed by FDG-PET scan. | Week 4, at the time of disease progression and 4 weeks after treatment is ceased.
The objective immune response as defined by achievement of a complete or partial response (irCR or irPR), based on irRECIST criteria. | End of week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Jayesh Desai, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Pham T, Pereira L, Roth S, Galletta L, Link E, Akhurst T, Solomon B, Michael M, Darcy P, Sampurno S, Heriot A, Ramsay R, Desai J. First-in-human phase I clinical trial of a combined immune modulatory approach using TetMYB vaccine and Anti-PD-1 antibody in patients with advanced solid cancer including colorectal or adenoid cystic carcinoma: The MYPHISMO study protocol (NCT03287427). Contemp Clin Trials Commun. 2019 Jul 10;16:100409. doi: 10.1016/j.conctc.2019.100409. eCollection 2019 Dec. PMID 31650066